CLINICAL TRIAL: NCT06829004
Title: Calf Circumference Adjusted for Body Composition to Assess Muscle Mass
Status: Not yet recruiting | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Alastair Forbes, Visiting Professor, University of Tartu
Other Study IDs: 396/T-16
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Muscle Mass; Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing bone density scanning at Tartu University Hospital: Patients undergoing bone density scanning at Tartu University Hospital selected from those attending the internal medicine clinics

SUMMARY:
Muscle mass is a critical indicator for malnutrition and sarcopenia assessment. Anthropometric measurements like calf circumference (CC) could be a simple and cost-effective alternative when gold standard methods are not available. However, CC is probably less accurate for estimating muscle mass in female patients and patients with obesity. This study investigates whether adjusting CC using mid-upper arm circumference (MUAC) improves muscle mass estimation in patients with obesity. If validated, this correction method would serve as a simple clinical tool for muscle mass assessment.

DETAILED DESCRIPTION:
The patient's demographic data including age, sex, primary diagnosis, and diagnoses of co-morbidities are found by the investigator in the medical history (eHL). The researcher codes the current main diagnosis and its severity: we use the World Health Organization's ICD-11 classification (icd.who.int/browse11/l-m/en) and a three-point scale where 1 is mild and 3 is severe.

The patient will be interviewed for changes in body weight and food intake. Anthropometric measurements will be recorded, including height, weight, body mass index (BMI), mid upper arm circumference, calf circumference, and waist circumference.

The accurate muscle mass measurement will be done using total body densitometry (DEXA) scan, that was already ordered for other purposes. Bone mineral density (BMD) from DEXA scan will be recorded. This allows us to see if calf circumference can be used for estimating bone mineral density. Patients will be followed up one year after data collection. Follow up will involve calling the patients and asking them questions from the SarQoL (sarcopenia quality of life questionnaire)

Calf circumference will be measured using non-elastic tape at the widest part of the dominant calf in the seated position with the weight evenly distributed on both feet (1). Mid upper arm circumference will be measured at the midpoint between the acromial surface of the scapula and the olecranon process of the elbow over the dominant arm when bent at 90 degrees. Waist circumference will be measured using measuring tape 2.5 cm above the umbilicus in a standing position. Waist circumference is used to define obesity as it is a marker of abdominal obesity (2). We aim to keep the interview no longer than 10 minutes.

Demographic and anthropometric data will be analyzed using descriptive statistics. The sensitivity, specificity of muscle mass measurements will be calculated. Corrected calf circumference will be compared to DEXA (gold standard diagnostic tool) and new cutoffs will be defined by using Receiver Operating Characteristic curves. Statistical analyses will be performed using R.

ELIGIBILITY:
Inclusion Criteria:

Booked to undergo bone density scanning (DEXA) at Tartu University Hospital

Exclusion Criteria:

Isolation for infectious disease Pregnancy and lactation Unable to understand or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the internal medicine clinic for whom diagnostic bone density scanning (DEXA) has been requested by the physician normally responsible for the patient's care
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of corrected calf circumference in estimating muscle mass | 15 months
  Accuracy of corrected calf circumference in estimating muscle mass in comparison to densitometry (DEXA) used as a gold standard

SECONDARY OUTCOMES:
Comparison of accuracy of corrected calf measurement results in female patients | 15 months
  Comparison of accuracy of results in female patients thought to be in greater need of correction
Comparison of accuracy of corrected calf measurement results in obese patients | 15 months
  Calf measurement results thought to be less reliable in obese patients
Quality of life with and without corrected results of anthropometry | 15 months
  Low muscle mass is associated with poor quality of life and may be estimated better with anthropometric corrections. Quality of life will be measured using the SarQoL tool designed to examine quality of life in sarcopenia (0-100 scale high being good)
Bone density estimated from corrected calf circumference | 15 months
  Bone density may be possible to estimate from corrected calf circumference

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, MD, Study Director — University of Tartu

IPD SHARING:
Plan to Share IPD: Undecided
Confidentiality issues prevent full access but we anticipate making anonymised data available to other investigators

REFERENCES:
- [Background] Deutz NEP, Ashurst I, Ballesteros MD, Bear DE, Cruz-Jentoft AJ, Genton L, Landi F, Laviano A, Norman K, Prado CM. The Underappreciated Role of Low Muscle Mass in the Management of Malnutrition. J Am Med Dir Assoc. 2019 Jan;20(1):22-27. doi: 10.1016/j.jamda.2018.11.021. PMID 30580819

DOCUMENTS (1):
  • Study Protocol (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT06829004/Prot_000.pdf